CLINICAL TRIAL: NCT03121417
Title: Biomarker-Driven Phase 2 Study of Nivolumab in Advanced Metastatic NSCLC
Brief Title: Nivolumab in Treating Patients With Advanced Metastatic Non-small Cell Lung Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Rathi Pillai, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00090380; NCI-2016-02017 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Winship3286-16-CA209-461 (Other: Emory University/Winship Cancer Institute)
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes on day 1. Courses repeat every 2 weeks in the absence of disease progression or unexpected toxicity
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab — 240 mg given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo

SUMMARY:
This phase II trial is studying blood and tumor tissue from patients with advanced non-small cell lung cancer who are treated with nivolumab to better understand how nivolumab works. Monoclonal antibodies, such as nivolumab, may interfere with the ability of tumor cells to grow and spread by turning on the immune system (T cells). We want to study the effects of nivolumab on the immune system (T cells) by collecting blood samples and samples from patients' tumors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To study the sustained proliferation of programmed cell death protein (PD)-1+Ki-67+cluster of differentiation(CD)8 T cells as a predictive biomarker of response to nivolumab by comparing the response rates to nivolumab treatment between two groups of patients (positive vs negative) stratified by the status of PD-1+Ki-67+CD8 T cells.

SECONDARY OBJECTIVES:

I. Characterize phenotype of proliferating T cells in peripheral blood in the setting of nivolumab therapy.

II. Perform gene expression profiling of activated T cells from peripheral blood.

III. Perform T cell receptor (TCR) sequencing of activated T cells from peripheral blood and tumor infiltrating T cells (TILs).

IV. Assess pre-treatment biopsies and biopsies at the time of disease progression for tumor infiltrating lymphocytes.

V. Determine progression free survival (PFS) and overall survival (OS).

OUTLINE:

Patients receive nivolumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 2 weeks in the absence of disease progression or unexpected toxicity.

After completion of study treatment, patients are followed up at 30 and 90 days and then every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed and dated an Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent form in accordance with regulatory and institutional guidelines; this must be obtained before the performance of any protocol related procedures that are not part of normal subject care
* Subjects must be willing and able to comply with scheduled visits, treatment schedule, laboratory tests, and other requirements of the study
* Histologically confirmed stage IV or recurrent non-small cell lung cancer (NSCLC) per the 7th International Association for the Study of Lung Cancer classification with squamous or non-squamous histology
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2; patients with PS 2 are being included as the primary endpoint of the study is correlation of blood based biomarkers with response; nivolumab is currently approved for both squamous and non-squamous NSCLC
* Disease progression following frontline platinum doublet therapy given for metastatic or recurrent disease; there is no restriction on prior lines of therapy following receipt of initial platinum doublet therapy

  * Continuation maintenance therapy following platinum-based chemotherapy will not be considered as a separate line of therapy
  * Prior platinum-containing adjuvant, neoadjuvant, or definitive chemoradiation therapy given for locally advanced disease is considered first-line platinum therapy only if recurrent disease developed within 6 months of completing therapy
  * Patients with activating epidermal growth factor receptor (EGFR) mutations must have received an EGFR tyrosine kinase inhibitor directed therapy prior to platinum therapy
  * Patients with anaplastic lymphoma kinase (ALK) translocations must have received an ALK tyrosine kinase inhibitor directed therapy prior to platinum therapy
* Prior systemic chemotherapy or other investigational therapy must have been completed at least two weeks prior to administration of nivolumab
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria
* Subject willing to undergo biopsy prior to treatment with investigational therapy for fresh tissue immune cell analysis and would consider biopsy at disease progression (progression biopsy is not mandated); biopsy should be obtained with core needle; fine needle aspirates are not sufficient; if prior archival tissue is available, it should be submitted
* Prior palliative radiotherapy must have been completed at least 2 weeks prior to registration; subjects with symptomatic tumor lesions at baseline that may require palliative radiotherapy within 4 weeks of randomization are strongly encouraged to receive palliative radiotherapy prior to randomization
* White blood cell (WBC) ≥ 2000/µL
* Neutrophils ≥ 1500/µL
* Platelets ≥ 100 x 10³/µL
* Hemoglobin > 9.0 g/dL
* Serum creatinine ≤ 2 x upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min (if using the Cockcroft-Gault formula)
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) ≤ 3 x ULN
* Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Women of childbearing potential (WOCBP) must use appropriate method(s) of contraception; WOCBP should use an adequate method to avoid pregnancy for 5 months (30 days plus the time required for nivolumab to undergo five half-lives) after the last dose of investigational drug
* Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab
* Women must not be breastfeeding
* Men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 7 months after the last dose of investigational product; women who are not of childbearing potential (i.e. who are postmenopausal or surgically sterile) as well as azoospermic men do not require contraception
* Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy; investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception; highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly
* At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as listed below:

  * HIGHLY EFFECTIVE METHODS OF CONTRACEPTION

    * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) by WOCBP subject or male subject's WOCBP partner
    * Nonhormonal IUDs
    * Tubal ligation
    * Vasectomy
    * Complete abstinence: Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs; subjects who choose complete abstinence are not required to use a second method of contraception, but female subjects must continue to have pregnancy tests; acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
  * LESS EFFECTIVE METHODS OF CONTRACEPTION

    * Diaphragm with spermicide
    * Cervical cap with spermicide
    * Vaginal sponge
    * Male condom without spermicide
    * Male condoms with spermicide
    * Progestin only pills by WOCBP subject or male subject's WOCBP partner
    * Female condom: A male and female condom must not be used together

Exclusion Criteria:

* Subjects with untreated central nervous system (CNS) metastases or carcinomatous meningitis are excluded
* Subjects with CNS metastases are only eligible if the CNS metastases are treated with radiotherapy and/or surgery and subjects are neurologically returned to baseline (except for residual signs or symptoms related to the CNS treatment); in addition, subjects must be either off corticosteroids, or on a stable or decreasing dose of ≤ 10 mg daily prednisone (or equivalent)
* Subjects must have recovered from the effects of major surgery or significant traumatic injury at least 14 days before registration
* Other active malignancy requiring concurrent intervention; a history of prior malignancy will not be an exclusion factor as long as the patient is not currently requiring treatment for this malignancy
* Subjects with an active, known or suspected autoimmune disease; subjects with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of registration; inhaled or topical steroids, and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of active autoimmune disease
* Subjects with interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected drug-related pulmonary toxicity
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-cytotoxic T-lymphocyte-associated protein (CTLA)-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection
* Ongoing or planned administration of anti-cancer therapies other than nivolumab
* Use of corticosteroids or other immunosuppressive medications per exclusion criteria
* Anti-cancer therapy, including an investigational agent, less than 14 days prior to the first dose of nivolumab
* Prisoners or subjects who are involuntarily incarcerated
* Any other serious or uncontrolled medical disorder, active infection, physical exam finding, laboratory finding, altered mental status, or psychiatric condition that, in the opinion of the investigator, would limit a subject's ability to comply with the study requirements, substantially increase risk to the subject, or impact the interpretability of study results
* Drugs with a predisposition to hepatoxicity should be used with caution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2019-03-09 (Actual); Study Completion 2019-03-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Up to 3 years after study start
  The response rates to nivolumab treatment will be compared between two groups of patients (positive vs negative) stratified by the status of PD-1+Ki-67+CD8 T cells. The objective disease response (ORR) is determined radiographically by Response Criteria in Solid Tumors version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Change in T cell population in the peripheral blood assessed by flow cytometry | Baseline up to 16 weeks after study start
  Fresh or frozen peripheral blood mononuclear cells (PBMCs) will be stained with anti-cluster of differentiation(CD)8, -CD4, -CD3, -CD45RA, -CC-chemokine receptor 7 (CCR7), -PD-1, -human leukocyte antigen(HLA)-antigen D related(DR), -CD38, -inducible co-stimulator(ICOS), -CD28, -CD27, -CD127, and -Tim-3. Live/Dead cell discrimination will be performed using fixable Dead Cell Stain Kit (Life Technologies). Samples will be acquired with LSR II flow cytometer (BD Biosciences) and analyzed using FlowJo software (Tree Star).
Progression Free Survival (PFS) | Every 12 weeks until disease progression or up to 3 years
  Patients will have tumor assessments per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 at 6 weeks (±1 week) following initiation of registration and treatment. Subsequent tumor assessments should occur every 6 weeks (±1 week) up to week 49, then every 12 weeks until disease progression. Patients will also have ongoing evaluation of peripheral blood immune cell populations and cytokines that will be analyzed and correlated with each restaging scan.
Overall survival (OS) | Every 3 months up to 3 years after drug discontinuation
  Patients who discontinue treatment with nivolumab on this protocol will be followed for survival follow-up data until death or conclusion of the study. They will be contacted every 3 months by telephone for survival follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Pillai, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University/Winship Cancer Institute, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/17/NCT03121417/ICF_000.pdf